CLINICAL TRIAL: NCT02101294
Title: Study Protocol for Carpal Tunnel Syndrome and Typing Keyboard: Controlled Randomized Trial
Brief Title: Study Protocol for CTS and Keyboard Controlled Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Finger Relief (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1997-01
Record Dates: First submitted 2014-03-24; First posted 2014-04-02 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel syndrome; repetitive stress disorder
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interossei Lumbricals Neuro Interface (Experimental): Comparison of report of symptoms of carpal tunnel syndrome when typing with standard QWERTY keyboard to report of symptoms of carpal tunnel syndrome when typing with Interossei Lumbricals Neuromuscular Technology Interface Therapy device.
  Interventions: Device: Interossei Lumbricals Neuro Interface; Device: Standard QWERTY keyboard

INTERVENTIONS:
Device: Interossei Lumbricals Neuro Interface — Finger Relief's keyboard home row layout [actual home row placement order: asdeihotlrn], plus substitutions on the upper row [qwfgjyuk;p] and bottom row [zxcvb'm,.] moves or shifts finger and thumb movement from the elbow muscles to the finger muscles. The movement of finger bending toward the palm is shifted to the interosseous and lumbrical muscles of the hand and fingers from the full flexion and extension muscle control to reduce contraction and expansion of tendons and the movement in the carpal canal adjacent to the median nerve and reduces pressure on the median nerve. Pressure on the median nerve compromises the nerve leading to symptoms of the carpal tunnel syndrome of pain, tingling, and numbness.
  Other Names: Finger Relief; Interossei Lumbricals Neuromuscular Technology Interface
Device: Standard QWERTY keyboard — Report of onset and severity symptoms of carpal tunnel syndrome when typing with QWERTY keyboard and the Finger Relief device.

SUMMARY:
The study hypothesis is that there is a relationship between the keyboard layout and carpal tunnel syndrome (CTS). Specifically, use of the standard QWERTY keyboard increases the risk of symptoms of carpal tunnel syndrome. The QWERTY keyboard requires more effort by the fingers than necessary to perform the required work, i.e. data or word entry; up to 200 percent more flexion and extension and 100 percent more distance traveled.

The purpose of the protocol is to evaluate two keyboard layouts for carpal tunnel syndrome therapy, and to see if the efficient keyboard, Finger Relief, can be used as an adjunctive tool to other treatments or therapy for CTS for typists. Subjects who had received a diagnosis of carpal tunnel syndrome from their medical doctor and, where not contraindicated, had received confirmation of the diagnosis of carpal tunnel syndrome with a nerve conduction velocity (NCV) study participated in four typing sessions to compare onset and severity of carpal tunnel symptoms. Testing sessions alternated between keyboards. The keyboard selected for the first typing session was determined by random assignment. Twenty subjects completed all four typing sessions. The test protocol consisted of a medical history, 3 tests of the subjective pain experience of the subject (visual analogue scale / verbal rating scale, and hand diagram), 2 clinical measures of physical manifestations of swelling associated with carpal tunnel syndrome (water volume/tape measure), and a measure of the length of time spent typing on each keyboard layout - QWERTY and TheOrdinals (the Finger Relief keyboard).

DETAILED DESCRIPTION:
The current study is the first clinical study of a keyboard with patients diagnosed with carpal tunnel syndrome. Previous research has compared the angular motion of the fingers in a comparison of QWERTY, Dvorak and Finger Relief keyboards (Robertson et al., 1995). However, in these studies the subjects had no diagnosis of carpal tunnel syndrome.

The typing test used typical English word combinations of letters which could be easily repeated for any layout. On the QWERTY keyboard, pressing the D and E flexes the middle finger. TheOrdinals letters (A D E H I L N O R S T) on QWERTY has 6 flexions, 1 each for the left middle; right middle, right ring, right index, 2 each left index fingers. TheOrdinals on Finger Relief keyboard have no flexions or extensions of the fingers The keystrokes were noted. The goal was to type to pain, change in feeling, numbness or tingling. The beginning and ending time was recorded manually with reference to a wristwatch or clock. Each of the four typing sessions ranged from 20 minutes (very little typing occurred) to more than an hour (extensive typing occurred without a report of symptoms). Pretyping measurement activities took about 10 minutes, including completing the analogue scaled self reporting test and water displacement test. Following this pretyping data collection, the subject was instructed to type until a change in pain was noticed. Post-typing measurement activities, including water displacement, a check for swelling, and self-report measures also took about 10 minutes.

The subject was then scheduled to return to the clinic no sooner than until an overnight had passed, or after any swelling has gone down. The protocol was repeated on a similar keyboard with only the letters rearranged. On the Finger Relief keyboard, pressing the D and E requires minimal flexion, as pressing the middle and index finger on the home row communicates the letters.

The study population was those who had been diagnosed with carpal tunnel syndrome. The FDA asked that the reference group consist of 20 individuals (no restrictions for the number of men and women). There were no minimum or maximum requirements of age, subjects were only required to have a history of carpal tunnel syndrome or similar problems when performing typing activities prior to study enrollment. Each subject confirmed a history of carpal tunnel syndrome, presumably causing difficulties in performing typing activities. However typing problems were not required for participation.

A total of 64 subjects responded to the study advertisements. Thirty-three of these subjects did not enter the study. Many were missing either the NCVS or a diagnosis of carpal tunnel syndrome from a doctor (14). Several did not respond to attempts to schedule study sessions (8). A few moved away from the area prior to study participation (4) or were too ill to participate (2). The remainder had insufficient interest to commit to participate in four testing sessions (3); were looking for treatment options, rather than a CTS study (1); or were advised by an attorney to decline participation in a CTS study, pending litigation that the subject was pursuing (1).

Thirty-one subjects completed the all steps before beginning the typing exercises, which included a medical history, informed consent, CTS diagnosis, and NCVS confirming the CTS diagnosis. Eleven withdrew or left the testing incomplete. Ten of the eleven dropouts were employed at office work, the other was employed as a registered nurse. Five withdrew prior to initiating study sessions. Six withdrew after beginning a study session but before completing the remaining sessions and did not respond to efforts to schedule the remaining tests. Four dropouts started with the QWERTY layout. Two started with Finger Relief. Four dropouts completed only one study session (three started with QWERTY, one began with Finger Relief). Two dropouts completed two study sessions (one began with QWERTY, one started with Finger Relief). Twenty subjects completed all 4 study sessions and are included in the analyses described in later sections of this application.

Swelling is a hallmark of CTS, because the median nerve must be compressed. Prior to this study, it was unknown whether swelling could be externally measurable in the least severe cases. Although the literature suggests that there is some swelling in all stages (1, 2 or 3) of CTS cases, the literature did not designate swelling by stage. Classic inflammation is measured by fever (rise in temperature), color (redness), swelling and pain. Only swelling and pain are externally measurable, without invasive procedures. The pre typing hand and wrist volume were the base line from which swelling was measured. Assuming typing causes measurable swelling, before the subsequent typing sessions, a sufficient time had to have passed for the swelling to return to base line. Thus, base line was defined as a return of external parameters (pain and swelling) to that which was measured before the first typing test session.

Swelling was measured by comparing the increase in hand volume before and after the activity as measured by the water displacement method. Water displacement was measured to determine if an increased amount of water from the hand and wrist measurement was displaced after typing on QWERTY keyboard as compared with typing on the TheOrdinals (the Finger Relief keyboard) keyboard. It was hypothesized that there would be a significant relationship between the increased amount of water and the use of the QWERTY keyboard.

The data were analyzed using a personal computer and statistical software. Calculations between the differences of means of swelling and pain, between the QWERTY and TheOrdinals (the Finger Relief keyboard) keyboards were completed. Regression techniques were used to estimate the differential impact of typing with each keyboard on swelling and pain. Means differences and regression techniques were also used to examine the effect of keyboard type on duration of typing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of carpal tunnel syndrome
* Completion of a nerve conduction velocity study (NCVS) within the past twelve months or a physician waiver of the NCVS
* Able to type using all fingers on the keyboard

Exclusion Criteria:

* Do not use all of their fingers when typing
* No active symptoms of carpal tunnel syndrome
* Unable to type, or flex and extend the fingers, for whatever reason
* Unable or unwilling to provide informed consent
* Use of pain relievers or medications during study sessions (potentially masking symptoms of median nerve entrapment)
* Unable to complete the typing activities before their symptoms (swelling associated with body ailments or metabolism) changed
* Had inconsistent subjective and objective evaluations in the preactivity test
* Threaten or abuse the investigator
* Unable to perform the activity so as to meet the minimal use requirements
* Had such injury as they had no sensation in their hands (i.e. Late stage)
* May suffer further injury (as indicated by their medical history) by attempting the typing activity
* Had non CTS related metabolic problems and upper extremity neurologic conditions, current or past, which have similar symptoms to median nerve entrapment, but which were not due to median nerve entrapment in the carpal canal

Ages: 12 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 1997-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John I Choate, J.D., Study Chair — Association of Repetitive Motion Syndromes
Locations (1):
- Finger Relief, Springfield, Virginia, United States

REFERENCES:
- [Background] Katz RT. Carpal tunnel syndrome: a practical review. Am Fam Physician. 1994 May 1;49(6):1371-9, 1385-6. PMID 7880220
- [Background] Endoscopic Carpal Tunnel Release by Chow in Arthroscopic Surgery, The Wrist, Whipple Ed. J. P. Lippincott Co. Philadelphia, 157 et seq
- [Background] CTS: relief at hand, School of Public Health, Vol. 11:4, UC Berkeley Wellness Letter, Jan. 1995, p. 7
- [Background] The Care of Minor Hand Injuries, Examination of the injured hand, p. 31-37, by Flatt, 4th ed. C.V. Mosby Com. St. Louis.
- [Background] Century of the Typewriter, by Beeching, Director, British Typewriter Museum, St. Martin's Press: New York, 1974, 28-43.
- [Background] 1994 Compton's Encyclopedia & fact-Index, Typewriter, at 342.
- [Background] Wood MB, Dobyns JH. Sports-related extraarticular wrist syndromes. Clin Orthop Relat Res. 1986 Jan;(202):93-102. PMID 3006958
- [Background] Kiefhaber TR, Stern PJ. Upper extremity tendinitis and overuse syndromes in the athlete. Clin Sports Med. 1992 Jan;11(1):39-55. PMID 1544186
- [Background] Weinstein SM, Herring SA. Nerve problems and compartment syndromes in the hand, wrist, and forearm. Clin Sports Med. 1992 Jan;11(1):161-88. PMID 1544180
- [Background] Van Handel PJ. The preparticipation fitness test. Clin Sports Med. 1991 Jan;10(1):1-18. PMID 2015635
- [Background] Herring SA, Nilson KL. Introduction to overuse injuries. Clin Sports Med. 1987 Apr;6(2):225-39. PMID 3319201
- [Background] Hunter SC, Poole RM. The chronically inflamed tendon. Clin Sports Med. 1987 Apr;6(2):371-88. PMID 3319206
- [Background] Common Hand Injuries and Infections, A practical approach to early treatment, by Carter, W. B Saunders, Co. Philadelphia et al, 1983, at pp. 170-175
- [Background] The Hand, Surgical and Non-surgical Treatment, by Kilgore and Graham, Lea & Febiger, Philadelphia, 1977.
- [Background] Carpal Tunnel Syndrome, The Johns Hopkins Medical Handbook, The 100 Major medical Disorders of People Over the Age of 50, by Margolis and Moses, Ed. The Johns Hopkins Medical Letter Health After 50, Rebus, New York, 382.
- [Background] Pigs, Ducks and RSI, Machrone, PC Magazine, May 17, 1994, v13 n9 p87(2).
- [Background] Neurology, Medical Library Lawyers Edition, by Ausman and Snyder, 6:105F, 1990.
- [Background] Carpal Tunnel Syndrome, in Rehabilitation, Medical Library Lawyers Edition, by Ausman and Snyder, 28:12, 1990.
- [Background] Joyce B, Moxley RA. August Dvorak (1894-1975): Early expressions of applied behavior analysis and precision teaching. Behav Anal. 1988 Spring;11(1):33-40. doi: 10.1007/BF03392452. PMID 22477993
- [Background] Hopkins A. The social recognition of repetition strain injuries: an Australian/American comparison. Soc Sci Med. 1990;30(3):365-72. doi: 10.1016/0277-9536(90)90191-t. PMID 2137940
- [Background] Gerriets JE, Curwin SL, Last JA. Tendon hypertrophy is associated with increased hydroxylation of nonhelical lysine residues at two specific cross-linking sites in type I collagen. J Biol Chem. 1993 Dec 5;268(34):25553-60. PMID 8244992
- [Background] Minami A, Ogino T, Tohyama H. Multiple ruptures of flexor tendons due to hypertrophic change at the distal radio-ulnar joint. A case report. J Bone Joint Surg Am. 1989 Feb;71(2):300-2. No abstract available. PMID 2918017
- [Background] Comparative Effects of QUERTY (sic) and DVORAK Keyboards in the NIOSH Health Hazard Evaluation at US West Communications, by Hales and Sauter, NIOSH, Cincinnati Ohio, circa 1995.
- [Background] Nerve Repair and Grafting, by Wilgis and Brushart, in Operative Hand Surgery, by Green Editor, 3d Edition, Vol. 2, Churchill Livingstone, New York, pp. 1315 et seq.
- [Background] Entrapment and Compression Neuropathies, by Eversmann, in Operative Hand Surgery, by Green Editor, 3d Edition, Vol. 2, Churchill Livingstone, New York, pp. 1346 et seq.
- [Background] Anto C, Aradhya P. Clinical diagnosis of peripheral nerve compression in the upper extremity. Orthop Clin North Am. 1996 Apr;27(2):227-36. PMID 8614575
- [Background] Kulick RG. Carpal tunnel syndrome. Orthop Clin North Am. 1996 Apr;27(2):345-54. PMID 8614583
- [Background] Mirza MA, King ET Jr. Newer techniques of carpal tunnel release. Orthop Clin North Am. 1996 Apr;27(2):355-71. PMID 8614584
- [Background] Einhorn N, Leddy JP. Pitfalls of endoscopic carpal tunnel release. Orthop Clin North Am. 1996 Apr;27(2):373-80. PMID 8614585
- [Background] Szabo RM, Madison M. Carpal tunnel syndrome. Orthop Clin North Am. 1992 Jan;23(1):103-9. PMID 1729659
- [Background] Essential elements of an upper extremity assessment battery, by Fess in Rehabilitation of the Hand Surgery and Therapy by Hunter et al Ed. 3d Ed. 1990, C.V. Mosby, St. Louis. 53 et seq. (splint and rehab forms)
- [Background] Clinical Examination of the Hand by Aulicino and DuPuy, in Rehabilitation of the Hand Surgery and Therapy by Hunter et al Ed. 3d Ed. 1990, C.V. Mosby, St. Louis. 31 et seq.
- [Background] Hunter JM, Mackin E. Management of edema. In: Hunter JM, ed. Rehabilitation of the Hand, Surgery and Therapy. 3rd ed. St Louis, Mo: CV Mosby Co; 1990:190-191.
- [Background] Nerve Lesions in Continuity by Spinner, in Rehabilitation of the Hand Surgery and Therapy by Hunter et al Ed. 3d Ed. 1990, C.V. Mosby, St. Louis. 523 et seq.
- [Background] Therapist's Management of carpal tunnel syndrome, by Baxter-Petralia, in Rehabilitation of the Hand Surgery and Therapy by Hunter et al Ed. 3d Ed. 1990, C.V. Mosby, St. Louis. 640 et seq. at 640.
- [Background] Carpal Tunnel Syndrome in Complete Guide to Sports Injuries by Griffith, at 380.
- [Background] Surgical and Diagnostic Procedures: Inappropriate Procedures: 1991 and 1992, Statistical Record of Health and Medicine, by Dorgan Ed. Gale Research, International Thomson Publishing, New York, 1995, p. 183, table 239.
- [Background] Carpal Tunnel Syndrome, Arm and Leg Surgery, The Surgery Book, 73 Most Common Operations, by Youngson, Diagram Group, St. Martins Press, 1993, p. 176 et seq.
- [Background] Pain in the hand and wrist. (ABC of Rheumatology) by Michael Shipley il v310 British Medical Journal Jan 28 '95 p239(5) Infotrac
- [Background] Lane, Merritt, Nathan: CTS: The workup. Patient Care Apr 15,1993, pp 97 108, Infotrac, management techniques, pp. 111, Kasdan, et al. Infotrac
- [Background] Sposato, Riley, Ballard, Stentz & Glisman v37 Jourl of Occupational & Environmental Medicine Sept '95 p1122(5)
- [Background] Franzblau A, Werner RA, Johnston E, Torrey S. Evaluation of current perception threshold testing as a screening procedure for carpal tunnel syndrome among industrial workers. J Occup Med. 1994 Sep;36(9):1015-21. PMID 7823213
- [Background] When to suspect - and diagnosis. (Carpal Tunnel Syndrome) by McCue and Mayer il v33 Consultant Dec '93 p40(4),
- [Background] Katz JN, Punnett L, Simmons BP, Fossel AH, Mooney N, Keller RB. Workers' compensation recipients with carpal tunnel syndrome: the validity of self-reported health measures. Am J Public Health. 1996 Jan;86(1):52-6. doi: 10.2105/ajph.86.1.52. PMID 8561242
- [Background] Relieve that tingling wrist! (caring for carpal tunnel syndrome)(includes related articles on causes of and how to avoid carpal tunnel syndrome) il v11 Health News Oct '93 p5(2)
- [Background] End of the tunnel. (using yoga to treat repetitive stress injuries) by Marty Munson v47 Prevention March '95 p22(2)
- [Background] Carpal tunnel syndrome protection. by Susan S. Lang v15 Computers in Libraries Feb '95 p10(2) copyright 1995 Meckler Corporation.
- [Background] Dissecting the CTS debate. (carpal tunnel syndrome) by Susannah Zak, Figura il v57 Occupational Hazards Nov '95 p28(4)
- [Background] A pain in the wrist. (repetitive strain injuries) (Backpack Healthwatch) by John DeMont il v107 Maclean's Nov 21 '94 p58(2)
- [Background] White KM, Congleton JJ, Huchingson RD, Koppa RJ, Pendleton OJ. Vibrometry testing for carpal tunnel syndrome: a longitudinal study of daily variations. Arch Phys Med Rehabil. 1994 Jan;75(1):25-8. PMID 8291957
- [Background] RSI suit turns into a legal pain for Apple. (repetitive strain injuries) (Brief Article) by Jon Swartz v9 MacWEEK March 6 '95 p22(2) copyright 1995 Ziff Davis Pub.
- [Background] A pain in the finger. (defining and preventing carpal tunnel syndrome) by Gordon Campbell v20 Computing Canada Oct 26 '94 p9(1), copyright 1994 Plesman Publications Ltd. (Canada).
- [Background] Vigorous defense stalls injury claims on repetitive strain. (repetitive strain injury case against IBM) by Steve Lohr 33 col in. v144 The New York Times May 29 '95 p19(N) pB7(L) col 6.
- [Background] IBM cleared in Nancy Urbanski Repetitive Strain Injury lawsuit) by Julie Pitta 14 col in. v114 Los Angeles Times March 9 '95 pD1 col 2.
- [Background] Flowers KR, McClure PW, McFadden C. Management of a patient with lacerations of the tendons of the extensor digitorum and extensor indicis muscles to the index finger. Phys Ther. 1996 Jan;76(1):61-6. doi: 10.1093/ptj/76.1.61. PMID 8545494
- [Background] Hamilton GF, Lachenbruch PA. Reliability of goniometers in assessing finger joint angle. Phys Ther. 1969 May;49(5):465-9. doi: 10.1093/ptj/49.5.465. No abstract available. PMID 5804302
- [Background] Quantification of Tendon Excursion through Kinematic Analysis of Typing Movements on Alternative Keyboard Layouts, by Flannery, of California State Univ. Sacramento, R. Robertson of Univ. of Pittsburgh Medical Center, and R. Cooper of Veterans Administration Hospital, in Conference Proceedings 19th Anual Meeting of the American Society of Biomechanics, Stanford University California, August 1995, pp.195-196.
- [Background] Neugebauer et al, Qualitative Meta Analysis in Principles and Practice of Research, Strategies for Surgical Investigators, 2d Ed. Troidl et al, Springer-Verlag, New York et al. p. 72-73.
- [Background] U.S. patent 5,352,050
- [Background] U.S. Patent 2,040,248 granted May 12, 1936.
- [Background] Wood-Dauphinee & Troidl, Ch. 17 Endpoints for Clinical Studies. pp. 151 et seq. Principles and Practice of Research. Strategies for Surgical Investigators, 2d ed. ed. by Troidl et al, Springer-Verlarg New York.
- [Background] Critical Appraisal of Published Research, pp. 7pp 84-85. Principles and Practice of Research, Strategies for Surgical Investigators, 2d ed. ed. by Troidl et al, Springer-Verlarg New York.
- [Background] Typing for everyone, by Levine, Arco Publishing, Inc, New York, 1980.
- [Background] Palmer DH, Hanrahan LP. Social and economic costs of carpal tunnel surgery. Instr Course Lect. 1995;44:167-72. PMID 7797856
- [Background] Silverstein BA: Fine LJ, ARmstrong TJ: Carpal tunnel syndrome: causes and a preventative strategy, Semin Occup Med 1:213-21, 1986.
- [Background] Armstrong TJ: An ergonomic guide to carpal tunnel syndrome, Akron, 1983, American Industrial Hygiene Association.
- [Background] Denys EH. AAEM minimonograph #14: The influence of temperature in clinical neurophysiology. Muscle Nerve. 1991 Sep;14(9):795-811. doi: 10.1002/mus.880140902. PMID 1656252
- [Background] Braun RM, Davidson K, Doehr S. Provocative testing in the diagnosis of dynamic carpal tunnel syndrome. J Hand Surg Am. 1989 Mar;14(2 Pt 1):195-7. doi: 10.1016/0363-5023(89)90005-1. PMID 2703665
- [Background] KENDALL D. Aetiology, diagnosis, and treatment of paraesthesiae in the hands. Br Med J. 1960 Dec 3;2(5213):1633-40. doi: 10.1136/bmj.2.5213.1633. No abstract available. PMID 13752458
- [Background] Typists' Speed & Efficiency, by Virginia Russell, Computer Technology Review, Winter 1985.
- [Background] Entrapment and Compression Neuropathies, by Eversmann, in Operative Hand Surgery, by Green Editor, 3d Edition, Vol. 2, Churchill Livingstone, New York, pp. 1346 et seq
- [Background] U.S. Pat. No. 5,718,590
- [Background] Blakiston's New Gould Medical Dictionary, copr. 1890-1956, McGraw-Hill Book Company, Inc. New York, Toronto, London; Editors Normand Hoerr, M. D., Arthur Osol, Ph.D. and 88 contributors.
- [Background] Dorland's Illustrated Medical Dictionary, 30th edition. 2003. Philadelphia Saunders. 22 Consultants. Anderson, Douglas Chief Lexicographer, Elsevier.
- [Background] Merriam-Webster http://www.merriam-webster.com/medical/ November 2009.
- [Background] www.cdc.gov/std/syphilis/STDFact-Syphilis.htm#symptoms centers for disease control and prevention

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Interossei Lumbricals Neuro Interface
Started | 31
Completed | 20
Not Completed | 11
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Population: Study participants had a physician diagnosis of carpal tunnel syndrome, confirmed with an abnormal result from a nerve conduction velocity study, and completed all 4 testing sessions.
Arm/Group | Interossei Lumbricals Neuro Interface
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 55 [18 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Length of Time Typing QWERTY Prior to Experiencing Symptoms of CTS (Carpal Tunnel Syndrome)
Description: Subjects were instructed to type until they experienced a change in symptoms, the length of time that the subjected typed until experiencing symptoms was recorded as this outcome measure. Length of time typing at each QWERTY session was averaged across the two sessions to determine Length of time typing QWERTY.
Time Frame: Participants will be assessed at each study of 4 sessions, two typing with the traditional QWERTY keyboard and two typing with the experimental device, each typing session will be separated by approximately one week to allow CTS symptoms to subside
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Length of Time Typing With QWERTY: Comparison of report of symptoms of carpal tunnel syndrome when typing with standard QWERTY keyboard to report of symptoms of carpal tunnel syndrome when typing with Interossei Lumbricals Neuromuscular Technology Interface Therapy device. These are the results of the length of time the patients typed with the QWERTY keyboard prior to stopping, averaged across two typing sessions.
Arm/Group | Length of Time Typing With QWERTY
Number analyzed (Participants) | 20
minutes | 71.063 (69.320)

2. Secondary Outcome: Measurement of Wrist Swelling Following Cessation of QWERTY Typing
Description: Before and after typing, the subject's wrists were measured with a tape measure. The change score is reported here.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters
Groups:
- Measurement of Wrist Swelling Following Typing With QWERTY: Comparison of report of symptoms of carpal tunnel syndrome when typing with standard QWERTY keyboard to report of symptoms of carpal tunnel syndrome when typing with Interossei Lumbricals Neuromuscular Technology Interface Therapy device. These are the results of the tape measurement of wrist swelling following typing with the QWERTY keyboard.
Arm/Group | Measurement of Wrist Swelling Following Typing With QWERTY
Number analyzed (Participants) | 20
centimeters | 0.560 (0.715)

3. Primary Outcome: Length of Time Typing FingerRelief Prior to Experiencing Symptoms of CTS
Description: Subjects were instructed to type until they experienced a change in symptoms, the length of time that the subjected typed until experiencing symptoms was recorded as this outcome measure, averaged across the two typing sessions that were FingerRelief.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Length of Time Typing With FingerRelief: Comparison of report of symptoms of carpal tunnel syndrome when typing with standard QWERTY keyboard to report of symptoms of carpal tunnel syndrome when typing with Interossei Lumbricals Neuromuscular Technology Interface Therapy device. These are the results of the length of time the patients typed with the FingerRelief keyboard prior to stopping, averaged across two typing sessions.
Arm/Group | Length of Time Typing With FingerRelief
Number analyzed (Participants) | 20
minutes | 98.35 (86.541)

4. Secondary Outcome: Measurement of Increase in Wrist Swelling Following FingerRelief Typing
Description: Before and after the typing session, the subject's wrist was measured. The mean change score of all participants is reported here.
Time Frame: Pre and Post
Measure: Mean (Standard Deviation); unit: centimeters
Groups:
- Measurement of Wrist Swelling Following FingerRelief: Comparison of report of symptoms of carpal tunnel syndrome when typing with standard QWERTY keyboard to report of symptoms of carpal tunnel syndrome when typing with Interossei Lumbricals Neuromuscular Technology Interface Therapy device. These are the results of the tape measurement of wrist swelling following typing with the FingerRelief keyboard.
Arm/Group | Measurement of Wrist Swelling Following FingerRelief
Number analyzed (Participants) | 20
centimeters | 0.042 (0.872)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at each typing session for the period of study data collection (1995-2008), over the course of thirteen years.
Description: No adverse events were recorded.
Arm/Group | Interossei Lumbricals Neuro Interface
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

LIMITATIONS AND CAVEATS:
Recruitment was a challenge and the budget to conduct the study was extremely limited. It took ten years to collect 20 participants who completed the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No